CLINICAL TRIAL: NCT03738826
Title: Reducing Disparities in Medication Adherence of Patients With Systemic Lupus Erythematosus (SLE)
Brief Title: Reducing Disparities in Medication Adherence in SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00100861; 5U54MD012530-02 (NIH)
Record Dates: First submitted 2018-11-06; First posted 2018-11-13 (Actual); Results first posted 2021-07-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Systemic Lupus Erythematosus
Keywords: medication adherence
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Medication Adherence | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Lupus clinic providers will use Surescripts refill information to assess adherence level and address adherence barriers. We will assess the feasibility and acceptability of the intervention.
  Interventions: Behavioral: Behavioral Intervention

INTERVENTIONS:
Behavioral: Behavioral Intervention — Lupus clinic providers will be prompted to assess adherence level using Surescripts refill information and address any adherence barriers that arise during the clinical encounter.

SUMMARY:
This is a pilot study to assess the feasibility of using Surescripts refill data during the clinical encounter to improve medication adherence in patients with systemic lupus erythematosus

ELIGIBILITY:
Inclusion Criteria

- All followup patients seen at the Duke Lupus clinic

Exclusion Criteria

* Patients not seen at the Duke Lupus Clinic
* New patients seen for the first time at the Duke Lupus Clinic
* Patients who are not prescribed any lupus medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai Sun, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun K, Eudy AM, Rogers JL, Criscione-Schreiber LG, Sadun RE, Doss J, Maheswaranathan M, Barr AC, Eder L, Corneli AL, Bosworth HB, Clowse MEB. Pilot Intervention to Improve Medication Adherence Among Patients With Systemic Lupus Erythematosus Using Pharmacy Refill Data. Arthritis Care Res (Hoboken). 2023 Mar;75(3):550-558. doi: 10.1002/acr.24806. Epub 2022 Nov 11. PMID 34739191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited over 12 clinic sessions between 9/25/19-1/25/20 from an academic lupus clinic, which takes place 1 half-day a week.
Groups:
- Lupus Clinic Providers: Lupus clinic providers will be prompted to assess adherence level using Surescripts refill information and address any adherence barriers that arise during the clinical encounter.
Period: Overall Study
Arm/Group | Behavioral Intervention | Lupus Clinic Providers
Started | 130 | 5
Completed | 130 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Intervention | Lupus Clinic Providers | Total
Number analyzed (Participants) | 130 | 5 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.0 (14.0) | 42.0 (4.9) | 43 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123 | 4 | 127
  Male | 7 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 127 | 5 | 132
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 71 | 0 | 71
  White | 54 | 4 | 58
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130 | 5 | 135

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Measured by Number of Participants With EMR (Electronic Medical Record) Documentation of Adherence
Description: Feasibility as measured by documentation of adherence assessment made by provider.
Time Frame: 12 weeks
Population: Data for this outcome measure collected on the Behavioral Intervention group only.
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Intervention | Lupus Clinic Providers
Number analyzed (Participants) | 130 | 0
Participants | 116 |

2. Primary Outcome: Acceptability as Measured by Provider Survey
Description: Acceptability as measured by provider survey, score range 1-5, with a higher score indicating that the intervention was more acceptable.
Time Frame: 12 weeks
Population: Data for this outcome measure collected on the Lupus Clinic Providers group only.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Behavioral Intervention | Lupus Clinic Providers
Number analyzed (Participants) | 0 | 5
score on a scale |  | 4.4 (0.6)

3. Secondary Outcome: Medication Adherence as Determined by Self Report
Time Frame: 12 weeks
Population: Data not collected.
Arm/Group | Behavioral Intervention | Lupus Clinic Providers
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Adherent Participants as Determined by Medication Possession Ratio (MPR)
Description: Medication Possession Ratio (MPR) = days with medication/total days. This will be determined by pharmacy refill data and calculated for 3 months (90 days). An MPR > or = 80% indicates adherence.
Time Frame: Baseline, 12 weeks
Population: Data for this outcome measure collected on the Behavioral Intervention group only.
Measure: Number; unit: percentage of participants
Arm/Group | Behavioral Intervention | Lupus Clinic Providers
Number analyzed (Participants) | 130 | 0
percentage of participants
  Baseline (prior to intervention) | 46 |
  12 weeks (after intervention) | 55 |

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Collected via chart review of clinic visit during which the intervention was performed.
Arm/Group | Behavioral Intervention | Lupus Clinic Providers
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/5
Other Adverse Events (participants affected / at risk) | 0/130 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-07): https://cdn.clinicaltrials.gov/large-docs/26/NCT03738826/Prot_SAP_000.pdf